CLINICAL TRIAL: NCT03230825
Title: Oral Contraceptive Pills Versus Expectant Management for Retained Pregnancy Products After a First Trimester Miscarriage: a Randomized Clinical Trial
Brief Title: Oral Contraceptive Pills Versus Expectant Management for Retained Pregnancy Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Anat Hershko Klement, Principal Investigator, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0263-16
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Retained Products of Conception Post Abortion
Keywords: incomplete abortion; retained products of conception; combined oral contraceptives; ultrasound
MeSH Terms: conditions — Abortion, Incomplete | interventions — Contraceptives, Oral; Watchful Waiting

STUDY DESIGN:
Intervention Model Description: Once informed consent forms are signed, the patient will be randomized (using a randomization table handled by a 3rd party) into one of 2 groups:
  1. Expectant management of 3 weeks and a follow up visit a week after.
  2. Oral contraceptive agent, given for free, for 3 weeks and a follow up visit a week after treatment withdrawal.
Who Masked: Outcomes Assessor
Masking Description: Data analysis will be performed according to group code .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral contraceptives (Experimental): Oral contraceptive agent, given for free, for 3 weeks and a follow up visit a week after treatment withdrawal.
  Interventions: Drug: Oral contraceptive
- Expectant management (Sham Comparator): Expectant management for 3 weeks and a follow up visit a week later.
  Interventions: Other: Expectant management

INTERVENTIONS:
Drug: Oral contraceptive — Daily oral contraceptive agent for 3 weeks (FLAME, containing 0.02 mg Ethinylestradiol and 0.075 mg Gestodene)
  Arms: Oral contraceptives
Other: Expectant management — No intervention and a follow up visit a wewk later
  Arms: Expectant management

SUMMARY:
We speculate that the use of combined oral contraceptives may be a possible solution to promote the management of retained pregnancy products versus expectant management. By withdrawing the pill, the endometrium is expected to shed in a synchronized fashion (estrogen and progestin withdrawal bleeding and may also shed the retained products of conception and avoid a surgical procedure with its related potential complications.

DETAILED DESCRIPTION:
Miscarriage is a common event in general gynaecological practice, and is an age-dependent outcome. It is estimated -that approximately 20 percent of clinically recognized pregnancies will result in a miscarriage, and the prevalence is much higher if preclinical pregnancies are included as well .Failure to pass the contents of the pregnancy is reported in 15% of patients going through a spontaneous 1st trimester miscarriage and a similar rate in patients going through an induced medical abortion after a spontaneous pregnancy loss (miscarriage) and planned pregnancy termination using PGE1 (MisWe speculate that the use of combined oral contraceptives may be a possible solution to promote the management of retained pregnancy products versus expectant management. The exposure to combined oral contraceptives is known to induce secretory and decidual changes in the endometrium .By withdrawing the pill, the endometrium is expected to shed in a synchronized fashion (estrogen and progestin withdrawal bleeding). We hypothesize that such withdrawal bleeding may also shed the retained products of conception and avoid a surgical procedure with its related potential complications. oprostol).

All patients diagnosed with RPOC according to the inclusion and exclusion criteria , will be asked to give their informed consent to take part in the study.

Once informed consent forms are signed, the patient will be randomized (using a randomization table handled by a 3rd party) into one of 2 groups:

1. Expectant management of 3 weeks and a follow up visit a week after.
2. Oral contraceptive agent, given for free, for 3 weeks and a follow up visit a week after treatment withdrawal.

We wish to emphasize that the current management in our ward is expectant management in the population eligible for this study.

All US scans will be performed by 2 qualified sonographers using a 7.5 MHz transvaginal transducer. 2D images in both sagittal and axial planes will be obtained. Sonographic features to be evaluated are: endometrial maximal thickness measured in the sagittal plan, presence or absence and size of an endometrial mass (3 dimensions) and grading of endometrial vascularity. Vascularity will be graded as type 0, 1, 2 or 3 defining no detectable, minimal (less then myometrium), moderate (nearly equal to myometrium) or marked vascularity respectively (4).

At enrollment the patient will be monitored and interviewed for the following variables :

Age, BMI, OB - GYN history, smoking status, Blood pressure, pulse rate,Temperature, blood count, HCG levels.

All patients will be invited to a follow up visit 3 weeks after randomization. The follow up visit will include again an ultrasound scan as described above.

In any case the patient is reporting a menstrual bleeding/ abdominal pain/ fever she will contact the 24hr available ER of the ward and will be evaluated for complications. After evaluation is completed the principal investigator will be contacted and the case will be discussed as for the need for additional measures and documented in the research file.

In the planned 4 week post randomization visit the following parameters will be monitored:

Blood pressure, pulse rate, Temperature, blood count, HCG levels as well as a review of any symptoms.

Following the interview a trans-vaginal scan will be performed in order to evaluate the cavity and any retained products existence and any presence of blood flow in case of a positive diagnosis.

In any case of retained products detected by ultrasound we will recommend a surgical hysteroscopy.

The oral contraceptives will be donated by DEXCEL LTD, ISRAEL to the hospital pharmacy, where it will be stored.

Brand name :FLAME containing 0.02 mg Ethinylestradiol and 0.075 mg Gestodene. Israeli authorities demand that a drug which is tested in a research will be provided to the participant without charging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients going through a Misoprostol or Misoprostol/Mifepristone induced procedure after a spontaneous 1st trimester pregnancy loss or as a 1st trimester planned pregnancy termination and present retained pregnancy products by a trans-vaginal ultrasound scan.
2. Patients after a surgical evacuation of pregnancy products (dilatation and curettage - D&C) of a 1st trimester miscarriage and present retained pregnancy products by a trans-vaginal ultrasound scan.
3. All retained products included are of a previously confirmed intra-uterine pregnancies.
4. Asymptomatic patients or mild symptoms of bleeding (spotting).
5. Presence of a measurable hyperechoic material by 2 dimensional TVUS

Exclusion Criteria:

1. Retained products with any of the following clinical presentations : more than a mild vaginal bleeding, hemodynamic instability, signs of infection and/or abdominal pain.
2. Any suspicion of a molar pregnancy.
3. A known contra-indication for the use of oral contraceptives

Ages: 16 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Retaiend pregnancy products
Enrollment: 100 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
persistent retained pregnancy products rate | 4 weeks
  rate

CONTACTS AND LOCATIONS:
Overall Officials: Anat Hershko Klement, MD, Principal Investigator — Meir Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen BA, Creinin MD. Medical management of early pregnancy failure: efficacy. Semin Reprod Med. 2008 Sep;26(5):411-22. doi: 10.1055/s-0028-1087107. Epub 2008 Sep 29. PMID 18825609
- [Background] Griebel CP, Halvorsen J, Golemon TB, Day AA. Management of spontaneous abortion. Am Fam Physician. 2005 Oct 1;72(7):1243-50. PMID 16225027
- [Background] Wang X, Chen C, Wang L, Chen D, Guang W, French J. Conception, early pregnancy loss, and time to clinical pregnancy: a population-based prospective study. Fertil Steril. 2003 Mar;79(3):577-84. doi: 10.1016/s0015-0282(02)04694-0. PMID 12620443
- [Background] Sellmyer MA, Desser TS, Maturen KE, Jeffrey RB Jr, Kamaya A. Physiologic, histologic, and imaging features of retained products of conception. Radiographics. 2013 May;33(3):781-96. doi: 10.1148/rg.333125177. PMID 23674774
- [Background] Casikar I, Lu C, Oates J, Bignardi T, Alhamdan D, Condous G. The use of power Doppler colour scoring to predict successful expectant management in women with an incomplete miscarriage. Hum Reprod. 2012 Mar;27(3):669-75. doi: 10.1093/humrep/der433. Epub 2012 Jan 9. PMID 22232130